CLINICAL TRIAL: NCT06802913
Title: A Novel Inhaled Formulation of Melatonin to Treat Adults With Insomnia Disorder: a Randomised Open-Label Crossover Trial
Brief Title: A Novel Inhaled Formulation of Melatonin to Treat Adults With Insomnia: Efficacy Study
Acronym: Mela-Nia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Hui Xin Ong, Dr, Woolcock Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18118
Record Dates: First submitted 2025-01-24; First posted 2025-01-31 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: Melatonin; Insomnia; Polysomnography; Biomarkers; Inhaled Therapy; Sleep Onset Latency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomised, open-label, crossover trial
Masking Description: As this trial is open-label, all study staff and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Melatonin Arm (Experimental): 100 µg daily of inhaled melatonin delivered by pressurized metered dose inhaler for two weeks before habitual bedtime.
  Interventions: Drug: Inhaled Melatonin (100 μg)
- Oral Melatonin Arm (Active Comparator): 4 mg daily of orally delivered melatonin tablets for two weeks before habitual bedtime.
  Interventions: Drug: Oral Melatonin (4 mg)

INTERVENTIONS:
Drug: Inhaled Melatonin (100 μg) — An orally inhaled formulation of melatonin delivered by pressurised metered dose inhaler (pMDI) to be taken before bedtime. The pMDI will deliver a total of 100 μg of inhaled melatonin (2 x 50 μg/actuation). The investigational product is produced under Good Manufacturing Practice by Ab Initio Pharma Pty Ltd, a GMP certified manufacturer of pharmaceutical products.
  Other Names: Melatonin
  Arms: Inhaled Melatonin Arm
Drug: Oral Melatonin (4 mg) — Two orally ingested tablets each containing 2 mg of melatonin (4 mg total) to be taken before bedtime. The investigational product is manufactured under Good Manufacturing Practice and is compliant with the TGA Therapeutic Order #101 that stipulates quality control requirements for capsule and pill-based products used in Australia.
  Other Names: N-Acetyl-5-methoxytryptamine; Circadin; Melatonin
  Arms: Oral Melatonin Arm

SUMMARY:
The goal of this clinical trial is to explore the potential benefits of an inhaled version of melatonin compared to oral melatonin tablets on adults with insomnia. The main question the trial aims to answer is: does inhaled melatonin affect the sleep profiles of adults with insomnia differently than oral melatonin tablets?

10 Participants will:

* Visit the research institute for a screening visit, for an overnight visit at the beginning of each study drug treatment and for a blood collection visit at the end of the conclusion of each study drug treatment period (5 visits in total)
* Take 100 µg of inhaled melatonin (2 inhaler puffs) nightly for two weeks
* Take a 4 mg of oral melatonin (2 tablets) nightly for two weeks

DETAILED DESCRIPTION:
This is a randomised open-label cross-over study of an inhaled formulation of melatonin (100 µg) versus oral melatonin tablets (4 mg) in adults with insomnia. The experiments performed for this trial will examine the effects of inhaled and oral melatonin on sleep microarchitecture such as sleep onset latency.

To be enrolled in the trial, participants are required to complete an online pre-screening survey. Eligible participants will be directed to a separate webpage where they will be invited to review and download the Participant Information Sheet (PIS) and asked to provide their contact details and consent for a follow up call/email from the research team to book in a screening visit. At the screening visit, the study team will explain the study to each participant and provide the opportunity to ask any questions. The study team will also ensure participants have had ample time prior to the visit to read and understand the PIS. The consent form will be signed by both the participant and a medical officer and participants. Once participants have joined the efficacy study, they will be randomised into their first treatment group; inhaled melatonin (100 µg) or oral melatonin tablets (4 mg).

Participants will attend the laboratory for an overnight visit then be treated with either inhaled melatonin or oral melatonin tablets before completing an overnight polysomnography sleep study. After the sleep study, participants will continue to take the study drug every night for two weeks and complete a sleep diary each morning to assess participant subjective perception of sleep quality. Once the two weeks of treatment have been completed, participants will visit the laboratory again to provide a blood sample that will be examined for biomarkers of neuroinflammation. There will be a 1 week washout period between treatment periods.

The study will recruit primarily through social media advertisements. The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Macquarie University, NSW, 2113, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia disorder as defined by the DSM-5 (difficulty initiating or maintaining sleep or waking up too early for at least 3 nights per week, for at least 3 months, with adequate opportunity and circumstances for sleep and at least one daytime impairment related to the sleep difficulty) and a score ≥15 on the ISI.
* History of subjective sleep onset latency (sSOL) ≥30 minutes on at least 3 nights per week in the previous 4 weeks.
* Able to provide informed electronic consent.
* Fluent English literacy.
* Adults aged 55+ years old.

Exclusion Criteria:

* People highly dependent on medical care as determined by a medical officer.
* Untreated moderate-severe sleep apnoea as diagnosed using in-home wrist oximetry (oxygen desaturation index>15, ongoing effectively treated sleep apnoea with insomnia will be allowed).
* Circadian disorders, narcolepsy, severe restless legs syndrome, and REM sleep behaviour disorder or uncontrolled psychiatric disorders.
* History of attempted suicide or current suicide ideation (indicated by a score >0 on Q9 of the Patient Health Questionnaire-9) at pre-screening.
* Objective cognitive decline measured by scoring ≤26 on the Montreal Cognitive Assessment (MoCA)
* Regular shift work, jet lag or trans-meridian travel (over 2h time difference) in the past week before randomisation.
* Pregnancy or lactation. Female participants of childbearing potential with a fertile sexual partner must have a negative serum pregnancy test result at the screening visit. Women will be advised to use contraception for the duration of the study.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical trial due to safety concerns or compliance with clinical study procedures.
* Currently participating in or has participated in a research study of an investigational agent or device within 4 weeks of enrolment.
* Ongoing use of anti-psychotic medication, bosentan, efavirenz, etravirine, modafinil, rifampin, carbamazepine or illicit stimulants.
* Regular use of hypnotics (including melatonin, valerian, kava, benzodiazepines and Z-drugs), and other medications that can cause additive sedation (e.g. sedating antihistamines, tricyclic antidepressants, antipsychotics) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Regular use of psychostimulants (e.g., dexamfetamine, lisdexamfetamine, methylphenidate) or non-amphetamine psychostimulants (e.g., armodafinil, modafinil, atomoxetine) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Use of antidepressant medications for treatment of low mood for less than one year or dose changes (escalation or tapering) or change in antidepressant medications within the past year.
* Regular use opioids within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Ongoing use of THC- or CBD-containing products within 14 days prior to the start of the trial.
* Dependence or any other drug or alcohol dependence within the past two years (alcohol to be limited to no more than 2 standard drinks per day during trial period).
* Regular use of drugs that are CYP1A2 inhibitors (e.g. amiodarone, cimetidine, ciprofloxacin, fluvoxamine) or CYP1A2 inducers (e.g. carbamazepine, phenobarbital, rifampin, tobacco).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sleep onset latency | Day 1
  Sleep onset latency (minutes) as assessed by polysomnography (PSG) on the first night of therapy. Sleep onset latency is the time between lights out and the first 30 second epoch scored as sleep using the American academy of sleep medicine criteria.

SECONDARY OUTCOMES:
Insomnia Severity Index | Measured during the initial screening visit and day 14 of treatment.
  The Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 28) regarding symptoms over the past 2 weeks. Scores range from 0-28 with higher scores indicating greater insomnia symptom severity.
Wake after sleep onset | Day 1
  Wake after sleep onset (WASO) is measured in minutes and is calculated from the first epoch of any sleep detected on the polysomnogram until the last epoch of sleep detected on the polysomnogram.
Total sleep time | Day 1
  Total sleep time (TST) is measured in minutes and is the sum of all 30 second epochs scored as sleep during an overnight polysomnogram.
Participant perception of sleep quality | Every observation for two weeks
  Ordinal rating of sleep quality (How would you rate the quality of your sleep? 9 = best ever sleep, 5 = neither best nor worst sleep, 1 = worst sleep ever), assessed in the Karolinska sleep diary after waking every day for two weeks.

OTHER OUTCOMES:
Traditional sleep staging | Day 1
  Proportion of the sleep opportunity scored at the 5 stages (wake, and N1, N2, N3, and REM sleep) between lights out and lights on, measured using overnight in-laboratory polysomnography, scored by a polysomnography technician in accordance with AASM Sleep Scoring criteria.
Absolute Electroencephalography (EEG) Power During Non-Rapid Eye Movement (NREM) Sleep | Day 1
  Spectral power of low delta (0.5-1 Hz), delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges between treatment arms. Power spectral analysis will be applied to EEG signals from polysomnography during NREM sleep after artefacts are detected and removed.
Absolute Electroencephalography (EEG) Power During Rapid Eye Movement (REM) Sleep | Day 1
  Spectral power of low delta (0.5-1 Hz), delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges between treatment arms. Power spectral analysis will be applied to EEG signals from polysomnography during REM sleep after artefacts are detected and removed.
Blood levels of glial fibrillary acidic protein | Day 14 of treatment.
  Blood-based glial fibrillary acidic protein (GFAP) within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of interleukin-6 | Day 14 of treatment.
  Blood-based interleukin-6 (IL-6), as measured by SIMOA blood neuro-metabolite assay.
Blood levels of plasma tau | Day 14 of treatment.
  Blood-based plasma tau within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of granulocyte-macrophage colony-stimulating factor | Day 14 of treatment.
  Blood-based granulocyte-macrophage colony-stimulating factor (GM-CSF) within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of brain derived neurotrophic factor | Day 14 of treatment.
  Blood-based brain derived neurotrophic factor (BDNF) within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of neurofilament light chain | Day 14 of treatment.
  Blood-based neurofilament light chain (NFL) within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of amyloid β (Aβ) | Day 14 of treatment.
  Blood-based Aβ (Aβ40:Aβ42 ratio) within each participant, as measured by SIMOA blood neuro-metabolite assay.
Blood levels of C-reactive protein | Day 14 of treatment.
  Blood-based C-reactive protein (CRP) within each participant, as measured by SIMOA blood neuro-metabolite assay.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Xin Ong, PhD, Principal Investigator — Woolcock Institute of Medical Research; Ron Grunstein, MBBS MD PhD FRACP, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon reasonable request to the Principal Investigators.
Time Frame: Non-identifiable IPD will become available one year after the Actual Study Completion Date and will remain available for fifteen years.
Access Criteria: Following Macquarie University access terms, access restrictions will be limited to appropriate permission, project proposal and approved from the investigator team and data custodian. Any Recipients of the data must obtain project and HREC approval prior to mediated access. The Coordinating Principal Investigator, Dr. Hui Xin Ong, will be retain access the de-identified data, stored on the Macquarie University Research Data Repository (RDR).
URL: https://libguides.mq.edu.au/research_data_repository